CLINICAL TRIAL: NCT06567067
Title: Human Factoring Validation Testing of the Pulsenmore ES Home Ultrasound Monitoring Device for Conducting Fetal Scans During Pregnancy
Brief Title: Human Factoring Validation of Pulsenmore ES Device
Status: Completed | Type: Observational
Sponsor: PulseNmore (Industry)
Responsible Party: Sponsor
Other Study IDs: SPRIM 22-1200
Record Dates: First submitted 2024-08-15; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Video guided: Participants will perform a scan using Pulsenmore ES device in the video mode independently following video tutorial. Participants will be remotely observed during the scan and interviewed by a human factoring researcher right after
  Interventions: Device: Pulsenmore ES home ultrasound
- Clinician guided: Participants will perform a scan using Pulsenmore ES device either in the clinician guided mode, guided by a health care professional via a telehealth visit. Participants and healthcare professionals will be remotely observed during the scan and interviewed by a human factoring researcher right after
  Interventions: Device: Pulsenmore ES home ultrasound

INTERVENTIONS:
Device: Pulsenmore ES home ultrasound — Fetal Ultrasound scanning using Pulsenmore ES device followed with an interview by a human factoring researched

SUMMARY:
The goal of this study is to conduct human factors validation testing with the Pulsenmore ES home Ultrasound device in the video-guided mode of operation (participants) and the clinician-guided mode of operation (participants and healthcare professionals (HCP)) to evaluate whether the device/user interface can be used by the intended users without any serious issues or errors under that intended use and actual use conditions. The intended users will be qualitatively assessed via observation and cognitive debrief and usability testing methodology. Participants will be remotely observed during the video-guided fetal scanning actual process and participants and HCPs will be remotely observed during the clinician-guided fetal scanning actual process.

ELIGIBILITY:
Inclusion Criteria for participants:

* The participant has voluntarily provided and signed the informed consent form (ICF)
* The participant has voluntarily provided authorization and signed the Videography and Photography Release form
* The participant is able to speak, read, write and comprehend US English and resides in the United States of America
* The participant to have adequate communications skills
* Pregnant women > 18 years of age
* A singleton gestation
* Gestational age between 14 to 38 weeks with a prior scan demonstrating fetal viability and confirming dates
* Maximum BMI of 40
* Willing and able to participate in a 60-75 min video and is willing to be audio recorded for the post-procedure interview

Inclusion criteria for HCP:

* The HCP has voluntarily provided and signed the HCP consent information sheet (CIS)
* The HCP has voluntarily provided authorization and signed the HCP Videography and photography Release form
* The HCP is able to speak, read, write and comprehend US English and resides in the United States of America.
* The HCP has adequate communications skills
* The HCP is willing and able to participate in one 60 min video call and is willing to be audio recorded during the interview.

Exclusion Criteria for participants:

* Multiple gestation
* Skin problem(s) in the abdominal area (such as wounds, cuts in the skin and skin rash)
* The participant has a visual or hearing impairment, and/or a condition that affects her motor and/or cognitive skills, that would prevent her from independently performing a fetal ultrasound scan at home
* The participant has a language barrier that can affect the communication and compliance to the usability study requirement
* Uncontrolled and untreated psychiatric conditions for a minimum of 6 months prior to screening,
* Alcohol or drug dependence with current symptoms
* Previous Pulsenmore ES trials and have previously used the Pulsenmore ES device
* Known fetal and genetic anomalies.

Exclusion criteria for clinicians:

* The HCP has a visual or hearing impairment, that would prevent him or her from independently directing a fetal ultrasound scan
* The HCP has a language barrier and/or in the opinion of the recruiting interviewer provides any reason to believe that compliance with the study requirements will not be achievable
* The HCP has participated in in previous Pulsenmore trials and have previously used the Pulsenmore ES device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants usability study will recruit singleton pregnant woman, gestational age (14-38 weeks) across al BMI groups and up to BMI 40.
  The healthcare professional (HCP) usability study will include only the first time the HCP performs the clinician-guided session.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Safety issues while using Pulsenmore ES device | One day
  Any safety issue, either serious that could cause serious injury or death to the user, or non serious
User error while using Pulsenmore ES device | One day
  Any user interface issues reported by study participants and HCPs that can cause delay in diagnosis or treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dallabrida, Principal Investigator — SPRIM PRO
Locations (2):
- United States (2):
  - Center for Fetal Medicine and Women Ultrasound, Los Angeles, California
  - Brigham and Women's Hospital, Boston, Massachusetts